CLINICAL TRIAL: NCT01554007
Title: Clinical Course of Crohn's Disease: a Prospective Multicenter Long-term Follow-up Study in Korea
Brief Title: Clinical Course of Korean Crohn's Disease Cohort
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Asan Medical Center (Other); Hanyang University (Other); Seoul National University (Other); Severance Hospital (Other); Samsung Medical Center (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Kyung Hee University Hospital at Gangdong (Other); Kangbuk Samsung Hospital (Other); Konyang University Hospital (Other); Korea University Anam Hospital (Other); Korea University (Other); Eulji General Hospital (Other); Eulji University (Other); SMG-SNU Boramae Medical Center (Other); Pusan National University Hospital (Other); Inje University (Other); Soonchunhyang University Hospital (Other); Songdo hospital (Unknown); Yeungnam University Hospital (Other); Wonkwang University (Other); Wonju Severance Christian Hospital (Other); Ewha Womans University (Other); Chonnam National University Hospital (Other); Jeju National University Hospital (Other); Chuncheon Sacred Heart Hospital (Other); Hangang Sacred Heart Hospital (Other); Dongtan Sacred Heart Hospital (Other); Chungbuk National University Hospital (Other); The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Associate Professor, Kyunghee University Medical Center
Other Study IDs: KCDC 2011-088
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease
MeSH Terms: conditions — Crohn Disease | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, DNA, and serum will be retained for central biobank
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Crohn's disease: Korean patients diagnosed with Crohn's disease
  Interventions: Other: Observation study

INTERVENTIONS:
Other: Observation study — No intervention was administered to the participants specifically for the purpose this study. Participant could be on any drug therapy.

SUMMARY:
In the past decade, the incidence and prevalence of CD (Crohn's disease) has continued to increase in Korea. Previous studies have indicated that Asian IBD (inflammatory bowel disease) patients differ from those of Western patients with regard to the genetic susceptibility and some clinical features. However, the available published data from retrospective studies in Korea were largely incomplete. The investigators aim of the study is a set-up of Korean cohort for CD, and thereby to assess the clinical course of Korean CD patients through a prospective multicenter long-term follow-up study. Secondary aims of this study are as follows: (1) to evaluate the efficacy, tolerability, and predictors to response to anti-TNF therapy for CD, (2) to identify the risk factors for postoperative recurrence on the basis of information obtained at initial diagnosis, and (3) to evaluate genotype-phenotype correlation.

DETAILED DESCRIPTION:
From 2009 to 2018, new cases of CD diagnosed will be recruited. Participants for this study will be enrolled from 33 academic teaching hospitals or colorectal specialized hospitals across Korea.

Medical records will be used to register demographic data, disease phenotype, the use of medication, flare-ups, surgery, hospitalizations, and mortality. Whole blood will be collected to central biobank with extraction of DNA ans seroum. The Montreal classification of Crohn's disease and the Crohn's disease activity index (CDAI) will be used to describe disease location, behavior and severity. F/U data will be analyzed using Kaplan-Meier analysis with log rank test and Cox regression analysis. An electronic database will be established in use of processing data.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 16
* Informed consent
* Patients who had a definitive diagnosis of Crohn's disease (documented by the standard clinical, radiographic, endoscopic, and histopathologic criteria)
* be capable of understanding the study and replying to the questionnaires

Exclusion Criteria:

* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: About 2000 patients diagnosed with Crohn's disease in the period of January 2009 to December 2018 in multiple hospitals in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To explore natural course of Crohn's disease and to identify prognostic factors for poor disease outcome in Korean patients with Crohn's disease | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Joo Sung Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (9):
- South Korea (9):
  - Hanyang University Guri Hospital, Guri-si
  - Kyunghee University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Chung-Ang University, Seoul
  - Inje University, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea St. Vincent Hospital, Seoul
  - Yonsei University; Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye BD, Yang SK, Cho YK, Park SH, Yang DH, Yoon SM, Kim KJ, Byeon JS, Myung SJ, Yu CS, Kim JH. Clinical features and long-term prognosis of Crohn's disease in Korea. Scand J Gastroenterol. 2010 Oct;45(10):1178-85. doi: 10.3109/00365521.2010.497936. PMID 20560811
- [Background] Kim ES, Kim WH. Inflammatory bowel disease in Korea: epidemiological, genomic, clinical, and therapeutic characteristics. Gut Liver. 2010 Mar;4(1):1-14. doi: 10.5009/gnl.2010.4.1.1. Epub 2010 Mar 25. PMID 20479907
- [Background] Ye BD, Jang BI, Jeen YT, Lee KM, Kim JS, Yang SK; IBD Study Group of the Korean Association of the Study of Intestinal Diseases. [Diagnostic guideline of Crohn's disease]. Korean J Gastroenterol. 2009 Mar;53(3):161-76. Korean. PMID 19835218